CLINICAL TRIAL: NCT04457661
Title: Evaluation of the Alcohol Elimination Effect of TCI711 Probiotic (Bacillus Coagulans) on Adult Individuals
Acronym: TCI711
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-036-A
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Breath Alcohol Level

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCI711 probiotic (Experimental): Taking one capsule (containing 10^10 of Bacillus coagulans TCI711) daily for one month
  Interventions: Dietary Supplement: Bacillus coagulans TCI711

INTERVENTIONS:
Dietary Supplement: Bacillus coagulans TCI711 — Using Bacillus coagulans TCI711 for one month and implementing alcohol testing at weeks 0, 1, and 4.

SUMMARY:
Investigating the possibility of using Bacillus coagulans TCI711 to improve the efficiency of alcohol removal in adult individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged between 20 to 60.
* Systolic pressure below 140
* Score of C-CAGE Questionnaire below 8 (male)/6 (female)
* Prohibiting other supplements before 2 weeks of the study and during the study
* Prohibiting alcohol drinks before 24 hours of the study
* Prohibiting caffeine drinks before 12 hours of the study

Exclusion Criteria:

* Alcohol or drug allergy
* Liver, kidney, cardiovascular, or chronic diseases
* Other severe disorders
* Hypertension
* Pregnancy or lactation
* Already involved in clinical testing
* Other supplements

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Breath Alcohol Level | 5 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.
Breath Alcohol Level | 15 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.
Breath Alcohol Level | 30 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.
Breath Alcohol Level | 60 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.
Breath Alcohol Level | 90 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.
Breath Alcohol Level | 120 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.
Breath Alcohol Level | 150 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.
Breath Alcohol Level | 180 minutes after drinking a certain volume of whisky
  A breathalyzer will be used for estimating blood alcohol content (BAC) from a breath sample.

CONTACTS AND LOCATIONS:
Locations (1):
- GeNext, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No